CLINICAL TRIAL: NCT06562387
Title: Transcranial Direct Current Stimulation (tDCS) as Adjunctive Therapy to Cognitive Stimulation in Medical Students With Depression
Brief Title: tDCS as Adjunctive Therapy to Cognitive Stimulation in Medical Students With Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Diana Guizar, Full-time tenured career professor, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FM/DI/56/2021
Record Dates: First submitted 2024-08-05; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Clinical Trial
Keywords: transcranial direct current stimulation; major depressive disorder; cognitive stimulation; Cognitive evoked potentials P300; cognitive impairment
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: single-blind, comparative clinical trial (cognitive stimulation + active tDCS vs. cognitive stimulation + sham tDCS). Randomization will be carried out with a list of numbers in Excel that will be in charge of one of the members of the research who will not have contact with the participants.
  The applicators of the stimulation techniques will be the same as those who evaluate and will not remain blind to the maneuver, unlike the students. All the applicators will be randomized to form the two groups and the applicator of the techniques will know whether it is the experimental maneuver or the placebo maneuver.
Who Masked: Participant, Care Provider
Masking Description: Regarding the simulated condition or sham, the equipment has the option inside to program it. It gives the options: Active / sham protocol, by default: ON - enables active stimulation and OFF - enables sham stimulation. The devices will be programmed, such that a few seconds of stimulation are administered at the beginning and end of the programmed time period to mimic the cutaneous perceptions (itching, tingling) that tend to be reported within the first moments of the stimulator being turned on, without being able to modify cortical excitability.
  The applicators of the stimulation techniques will be the same as those who evaluate and will not remain blind to the maneuver, unlike the students. All the applicators will be randomized to form the two groups and the applicator of the techniques will know whether it is the experimental maneuver or the placebo maneuver.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1. tDCS active (Active Comparator): Cognitive Stimulation + tDCS active in the Dorsolateral Prefrontal Cortex (Dorsolateral Prefrontal Cortex) to improve scores on tests of cognitive functioning (attention, memory, coordination, perception, reasoning and processing speed) and P300 cognitive evoked potentials.
  Interventions: Device: transcranial direct current stimulation; Other: cognitive stimulation
- 2. sham tDCS (Sham Comparator): Cognitive Stimulation + sham tDCS in the Dorsolateral Prefrontal Cortex (Dorsolateral Prefrontal Cortex) to improve scores on cognitive functioning tests (attention, memory, coordination, perception, reasoning and processing speed), and evoked potentials P300
  Interventions: Other: cognitive stimulation; Device: sham transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation is one of the most studied techniques in noninvasive neuromodulation. With a very good safety profile and low cost, it has been widely used to modulate cognition and behavior in both experimental and clinical settings. A growing body of literature, including randomized controlled trials, reports the clinical benefits of tDCS for many psychiatric symptoms, such as depression, anxiety, psychosis, addiction, and cognitive functions. tDCS has considerable potential as a treatment due to its relative cost, portability, safety, and ease of use compared to other neuromodulation methods. Early studies evaluated the effects of tDCS on the motor cortex; however, more recent research has also focused on its effects on the dorsolateral prefrontal cortex (DLPFC), in particular for treating psychiatric disorders and modulating cognitive performance.
  Arms: 1. tDCS active
Other: cognitive stimulation — This brain stimulation program is based on cognitive reserve and neuronal plasticity to improve mental performance through online games. The activities presented in this tool combine different therapeutic exercises, rehabilitation and learning techniques aimed at retraining and improving the skills most needed by each person. The intervention battery has multi-disciplinary tasks organized in a systematic and strategic way. To make these materials accessible, they are presented in the form of simple games that can be easily practiced through any computer or device. These cognitive stimulation tools are aimed at both healthy subjects and people concerned about their brain health, or patients with some kind of injury or decline in the central nervous system.
Device: sham transcranial direct current stimulation — Regarding the simulated condition or sham, the equipment has the option inside to program it. It gives the options: Active / sham protocol, by default: ON - enables active stimulation and OFF - enables sham stimulation. The devices will be programmed, such that a few seconds of stimulation are administered at the beginning and end of the programmed time period to mimic the cutaneous perceptions (itching, tingling) that tend to be reported within the first few moments of stimulator on, without being able to modify cortical excitability.
  Arms: 2. sham tDCS

SUMMARY:
Major depressive disorder (MDD) is a major public health problem, it negatively affects cognition and cognitive deficits affect information processing speed, attention, memory, executive function and working memory. In addition, cognitive deficits associated with MDD do not resolve after successful treatment of depressive symptoms. In one study, 94% of individuals with MDD and cognitive deficits at the start of treatment retained these deficits one year later, despite achieving clinical remission. Long-term maintenance of antidepressants does not prevent cognition decline, despite maintaining recovery from depression. Cognitive stimulation, has shown the potential to produce broad benefits primarily in working memory. The anodal tDCS increases task-related CPFdl activation. Furthermore, anodal tDCS on CPFdl has been shown to facilitate working memory processes, making tDCS a promising tool for the amelioration of depression-induced working memory impairment in a population with a high prevalence of depression and/or stress, such as medical school students.

Research question: Is Cognitive Stimulation (CS) + active tDCS in CPFdl more effective compared to sham CS+ tDCS in improving on working memory test scores, cognitive functioning, P300 cognitive evoked potentials and academic performance in medical students with depressive symptomatology? Aims: To evaluate the effect of active CE + tDCS in CPFdl to improve scores on tests of working memory, cognitive functioning, P300 cognitive evoked potentials and academic performance in medical students with depressive symptomatology vs sham CE + tDCS.

Materials and Methods: This is a single-blind, comparative (cognitive stimulation + active tDCS vs cognitive stimulation + simulated tDCS), randomized, longitudinal and prolective clinical trial. Analysis: A descriptive analysis of demographic and clinical characteristics will be performed with frequencies and percentages for categorical variables and with means and standard deviations for dimensional variables. Mean comparison tests (t-tests), analysis of variance (ANOVA) and correlation tests. Significance level p≤0.05.

DETAILED DESCRIPTION:
Cognitive training has demonstrated the potential to produce broad benefits in functional cognitive. As a fundamental and essential cognitive skill and essential, working memory supports complex thinking, but has limited capacity. Therefore, working memory training interventions have become popular as a means of potentially improve cognitive skills related to working memory for those who need it (Au et al.,2016) Transcranial direct current stimulation is one of the most widely studied techniques in neuromodulation non-invasive neuromodulation. With a very good safety profile and low cost, it has been widely used to modulate cognition and behavior in both experimental and clinical settings A growing body of literature, including randomized controlled trials, reports the clinical benefits of tDCS for many clinical benefits of tDCS for many psychiatric symptoms, such as depression, anxiety, psychosis, addiction, and cognitive function. tDCS has considerable potential as a treatment because of its relative cost, portability, safety, and ease of use compared with other neuromodulation methods. Early studies evaluated the effects of tDCS on the motor cortex; although more recent research has also focused on its effects on the dorsolateral prefrontal cortex (DLPFC), particularly for treating psychiatric disorders and modulating cognitive performance.

Side effects, such as itching, burning sensation or headache are common, but generally mild and without long-term impact.

Therefore, tDCS compares favorably with other therapeutic approaches such as antidepressants or transcranial magnetic simulation (TMS).

Transcranial direct current stimulation (tDCS), which has shown potential to modulate cortical excitability and cortical activity of the brain, by transmitting a weak electrical current to the brain, has been found as a possible way to improve working memory, sustained attention, motor learning, multitasking. Therefore, cognitive enhancement through tDCS has attracted increased attention over the last decade. A considerable number of single-session studies using tDCS have studies using tDCS have revealed potential benefits for improving participants' performance on working memory tasks. In a particularly anodal tDCS (a-tDCS) applied to the left dorsolateral prefrontal cortex, increased accuracy of response of the working memory task performed at the same time as the stimulation. However, no significant effect appeared when they applied anodal stimulation to the primary motor cortex and cathodal stimulation to the primary motor cortex and cathodal stimulation on the left CPFdl. These findings indicate that the potentiating effect of tDCS on working memory recall depends on the polarity of stimulation and is specific to the site of stimulation . Many subsequent studies compared factors such as electrode placement electrode placement, current density, and duration of stimulation that may affect the efficacy of tDCS and found that anodal stimulation of the left prefrontal tended to improve MT performance. Neuroimaging studies utilizing EEG and functional near-infrared spectroscopy (fNIRS) have provided evidence that tDCS may alter brain activities. In addition to studies related to working memory, tDCS has also shown potential to mitigate decreased vigilance and improve multitasking performance.

Based on the assumption that tDCS has the potential to modulate neuronal excitability and synaptic plasticity, several studies have explored the effect of tDCS on training cognitive training in the last 3 years. One study in a non-human primate model found that tDCS, together with multi-session learning, facilitated associative learning and altered functional connectivity when analyzing behavioral outcomes and local field potential. In a study of three-session working memory training, implemented in healthy adults, the advantage of working memory training combined with a working memory training combined with a-tDCS was not only present immediately following training, but also in the follow-up session up to 9 months after training. The benefits related to A-tDCS remained stable even up to one year after the original intervention, in a study of working memory training paired with 7-day tDCS in healthy young adults. Improved cortical efficiency and connectivity was also demonstrated in a study that found a significant improvement in cortical working memory through working memory training paired to -tDCS in healthy young adults.

A recent study in monkeys provided evidence that single-neuron activation rates and network interactions could be be modulated by polarity, and a dose of tDCS and a higher intensity of a-tDCS induced higher activation rates of regularly firing neurons. Although some reviews questioned the efficacy of tDCS, these recently published studies provide further evidence that working memory training combined with tDCS working memory training combined with tDCS can enhance cognition.

Patients with depression exhibit cognitive deficits in several domains (i.e., psychomotor speed, executive functions, memory, and attention), factors such as severity of depression are associated with greater cognitive deficits and lower remission rates, even after antidepressant treatment. These issues highlight the importance of investigating cognitive deficits in major depressive disorder.

However, only a few studies have investigated the brain mechanism underlying the effects of tDCS on cognition effects of tDCS on cognitive processing, with P300. Thus, the present project contributes in to propose a new treatment alternative for cognitive symptoms in MDD, to assist the pharmacological treatment, in addition to an early detection in terms of prevention of cognitive deterioration, providing new cognitive impairment, providing new tools for the diagnostic approach and management of this entity.

HYPOTHESIS Personalized cognitive stimulation in conjunction with transcranial direct current stimulation tDCS will be more effective compared to personalized cognitive stimulation + tDCS-placebo or sham in improving scores on neuropsychological neuropsychological test scores on the cognitive variables to be studied, cognitive potentials P300 and academic performance in UNAM medical students with depressive symptoms at 15 treatment sessions (acute phase) and at 15 sessions of treatment (acute phase) and at 4 weeks of maintenance.

After cognitive stimulation and tDCS, it is expected that in the experimental group the amplitude will be greater in the P300 component since the P300 component ncreased mastery of attention and working memory processes.

ELIGIBILITY:
Inclusion Criteria:

1. Age18 - 30 years old.
2. Vaccinated against SARS-COV2 virus.
3. Students of the Faculty of Medicine of the UNAM.
4. Fluent in Spanish.
5. Adequate visual and auditory acuity to be able to perform neuropsychological tests and perform cognitive stimulation.
6. Depressive symptoms with working memory impairment (diagnosed by applying a specific neuropsychological battery).
7. That they are not under antidepressant pharmacological treatment prior to admission to the research.
8. Good general health without medical illnesses (systemic arterial hypertension, diabetes mellitus, dyslipidemias, infections, thyroid disease, vitamin deficiencies) that do not interfere with the study.
9. Willingness to participate in a scheduled 8-week study and able to attend scheduled evaluations.

Exclusion Criteria:

1. Any neurological disease that allows suspicion of cognitive failure other than depression, such as Parkinson's disease, multiple infarct dementia, Huntington's disease, hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, history of head injury with loss of alertness.
2. Participants with history with severe psychiatric disorders according to DSM-5 (bipolar disorder, schizophrenia, chronic depression) or psychotic features, agitation or behavioral problems in the last three months that could lead to difficulties in complying with the protocol.
3. History of psychoactive substance abuse and current alcohol use with pattern of abuse or dependence in the past two years.
4. Participants with alterations in a conventional electroencephalogram (paroxysmal phenomena identified by a neurophysiologist).
5. Participants with pacemakers, intracranial metal objects or history of brain surgery, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2025-08-26 (Estimated)

PRIMARY OUTCOMES:
To compare performance on Cognitive improvement (Montreal Cognitive Assessment) between active and sham tDCS groups | three months
  remain the same or increase by 1 point on the Montreal Cognitive Assessment. MoCa assesses seven areas of cognition for a total possible score of 30 points. A score of 25 or less is indicative of cognitive impairment.
To compare performance on neuropsychological battery between active and sham tDCS groups | three months
  To compare performance on neuropsychological battery (Brief Visuospatial Memory Test, Stroop color test, Stroop color-word test, Trail Making Test-Part A and Part B, Verbal Learning Memory Test, Wisconsin Card Sorting Test, Weschler Memory Scale) between active and sham tDCS groups. To assess global cognition at each time point, we calculated a composite score by averaging the Z scores from these outcome measures. The mean and SD of the baseline scores were used to calculate Z scores both at baseline and at follow up time points.

SECONDARY OUTCOMES:
To compare Electrophysiological improvement on P300 between active and sham tDCS groups | three months
  increase P300 amplitude from the seventh stimulus onwards *p>0.05

OTHER OUTCOMES:
Global improvement or response to treatment | six months
  remain the same or have increased 1 point on the Clinical Global Impression Scale. The higher the score, the better the overall performance.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Patricia Guízar Sánchez, PhD, Principal Investigator — Universidad Nacional Autonoma de Mexico
Locations (1):
- Universidad Nacional Autónoma de México, Mexico City, Coyoacan, Mexico

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participan data available

REFERENCES:
- [Background] Begemann MJ, Brand BA, Curcic-Blake B, Aleman A, Sommer IE. Efficacy of non-invasive brain stimulation on cognitive functioning in brain disorders: a meta-analysis. Psychol Med. 2020 Nov;50(15):2465-2486. doi: 10.1017/S0033291720003670. Epub 2020 Oct 19. PMID 33070785
- [Background] Chase HW, Boudewyn MA, Carter CS, Phillips ML. Transcranial direct current stimulation: a roadmap for research, from mechanism of action to clinical implementation. Mol Psychiatry. 2020 Feb;25(2):397-407. doi: 10.1038/s41380-019-0499-9. Epub 2019 Aug 27. PMID 31455860
- [Background] Jog MV, Wang DJJ, Narr KL. A review of transcranial direct current stimulation (tDCS) for the individualized treatment of depressive symptoms. Pers Med Psychiatry. 2019 Nov-Dec;17-18:17-22. doi: 10.1016/j.pmip.2019.03.001. Epub 2019 May 7. PMID 31938757
- [Background] Jin J, Al-Shamali HF, McWeeny R, Sawalha J, Shalaby R, Marshall T, Greenshaw AJ, Cao B, Zhang Y, Demas M, Dursun SM, Dennett L, Suleman R. Effects of Transcranial Direct Current Stimulation on Cognitive Deficits in Depression: A Systematic Review. Psychiatry Clin Psychopharmacol. 2023 Dec 1;33(4):330-343. doi: 10.5152/pcp.2023.22583. eCollection 2023 Dec. PMID 38765850

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT06562387/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT06562387/ICF_001.pdf